CLINICAL TRIAL: NCT07084389
Title: A Financial Social Work Intervention for Families With Complex Financial Difficulties - A Randomised Controlled Trial
Brief Title: A Financial Social Work Intervention for Families With Complex Financial Difficulties (FinSoc)
Acronym: FinSoc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Anniina Kaittila, university lecturer, associate professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FinSoc; VN/10969/2024 (Other: Ministry of Social Affairs and Health Finland)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Financial Difficulties
Keywords: financial difficulties; social work; poverty; financial literacy; economic self-efficacy; financial anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: FinSoc intervention (Experimental): FinSoc intervention FinSoc intervention is delivered to the Experimental group by their social worker or social work professional.
  Interventions: Behavioral: FinSoc
- FinSoc control group (No Intervention): No Intervention: Control The control group will receive the usual social work services. After the third measurement point, they will receive a materials package.

INTERVENTIONS:
Behavioral: FinSoc — Financial Social Work intervention (FinSoc) The FinSoc intervention is a structured financial social work program designed for families experiencing complex financial difficulties. It consists of five modules, each delivered in a one-on-one session with a trained social worker. The modules focus on key areas such as budgeting, emotional and relational aspects of money, financial decision making, building long-term financial capability. The intervention aims to reduce financial anxiety, strengthen economic self-efficacy, and support overall wellbeing. Motivational interviewing techniques and client-centred approaches are used throughout to encourage active participation and goal-setting.
  Arms: Experimental: FinSoc intervention

SUMMARY:
As of 2022, about 12% of children in Finland lived in poverty. Many of these families face not only a lack of money but also stress, low confidence in managing finances, and limited access to financial guidance. This study aims to support these families by improving their financial skills and well-being through a practical and research-based program.

As of 2022, about 12% of children in Finland lived in poverty. These families often face not only financial hardship but also stress, low confidence in managing money, and limited access to financial guidance. The FinSoc study supports such families by improving financial skills and well-being through a practical, research-based program.

The intervention includes five sessions with a trained social service professional, focusing on budgeting, financial decision-making, emotions around money, and the role of money in relationships. The goal is to reduce financial anxiety, improve knowledge, and build confidence in managing finances. The sessions also aim to help families talk more openly about money and set realistic financial goals.

To test effectiveness, a randomized controlled trial (RCT) will be conducted. Families are randomly assigned to either the intervention group (receiving the FinSoc program) or a control group (receiving regular social work services and, after final measurements, a material package to promote financial capability).

At least 88 participants-families with at least one child under 18 and facing financial difficulties-will take part. Information will be collected at three time points: before the intervention, after it ends, and three months later. Outcomes include financial literacy, financial anxiety, economic self-efficacy, and health-related quality of life, measured with self-rating scales in questionnaires.

In addition to questionnaires, interviews will be conducted with a sample of families and social workers to explore their experiences-what worked, what could be improved, and how the sessions were received. This qualitative feedback will guide future development.

Formative evaluation involves feedback from families before and after each session, covering topic clarity, session usefulness, and experiences with the techniques. For fidelity assessment, social workers will report after each session on adherence to the planned approach and tool use.

The FinSoc program is offered through public and private social service providers. It was developed and is being implemented by an interdisciplinary team with expertise in financial social work, social policy, and mental health.

The study aims to improve families' everyday lives, inform social work practices, and contribute to knowledge on social and economic well-being.

ELIGIBILITY:
Inclusion Criteria:

* Client status in child welfare services, family social work, or adult social work
* Within the past six months, the client has brought up one or more of the following challenges in managing their finances during their contact with social services: (1) Difficulties paying bills, housing-related expenses, or repaying debts on time, (2) Difficulties meeting the basic needs of family members (e.g. food, medication, clothing) (3) A perceived lack of sufficient knowledge, skills, or competence to manage financial matters (4) Feelings of anxiety or stress related to financial situation.
* There is at least one underage child in the family. In cases of shared custody, the child must reside in the household for an average of at least half of the time in each calendar month.

Exclusion Criteria:

* There is an ongoing crisis or life situation in the family that, in the assessment of the social worker, prevents commitment to the intervention process.
* There is an active criminal proceeding within the family.
* The parents do not speak Finnish (all project materials are in Finnish, and there are no resources available to provide translations into other languages).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Financial Literacy Scale | Measured at three timepoints: 1) baseline pre-randomization, 2) within 1 week post-intervention for intervention group and at 3 months post-baseline for control group, 3) 3 months after previous measurement
  The primary outcome variable, financial literacy, is measured using an adapted version of the Financial Literacy Questionnaire developed by the Organisation for Economic Co-operation and Development (OECD). In this study, only items related to financial behaviour are included. Financial literacy is thus assessed using four statements: (1) 'Before I buy something, I carefully consider whether I can afford it'; (2) 'I pay my bills on time'; (3) 'I keep a close personal watch on my financial affairs'; and (4) 'I set long-term financial goals and strive to achieve them.' Each item is rated on a five-point Likert scale from 1 (completely disagree) to 5 (completely agree). The total score ranges from 4 to 20, with higher scores indicating greater financial literacy.

SECONDARY OUTCOMES:
Economic Self-Efficacy | Measured at three timepoints: 1) baseline pre-randomization, 2) within 1 week post-intervention for intervention group and at 3 months post-baseline for control group, 3) 3 months after previous measurement.
  Economic self-efficacy is measured using the Scale of Economic Self-Efficacy, which consists of ten items rated on a five-point Likert scale from 1 (completely disagree) to 5 (completely agree). The total score ranges from 10 to 50, with higher scores indicating greater economic self-efficacy.
Financial Anxiety | Measured at three timepoints: 1) baseline pre randomization, 2) within 1 week post-intervention for intervention group and at 3 months post-baseline for control group, 3) 3 months after previous measurement.
  Financial anxiety is assessed using the Financial Anxiety Scale (FAS), which consists of eight items rated on a four-point Likert scale ranging from 1 (totally untrue) to 4 (totally true). The total score ranges from 8 to 32, with higher scores indicating greater financial anxiety.
Health related quality of life | Measured at three timepoints: 1) baseline pre-randomization, 2) within 1 week post-intervention for intervention group and at 3 months post-baseline for control group, 3) 3 months after previous measurement
  Health-related quality of life is measured using the full Health-related quality of life is measured using the full Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale (11 items; PROMIS Global Health v1.2). The scale includes six items scored from 1 (poor) to 5 (excellent), with a total possible raw score range of 6 to 30; three items with question-specific 1-5 scales, yielding a combined score range of 3 to 15, where higher scores reflect better health; and one item assessing pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain). Thus, higher scores on the first nine items indicate better outcomes, while the pain item is reverse-coded so that higher values represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anniina Kaittila senior lecturer, PhD, Study Director — University of Turku
Locations (1):
- Univeristy of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
The data is sensitive and must not be shared outside of the research group.

REFERENCES:
- [Background] OECD INEF. (2018). Organisation for Economic Co-Operation and Development. OECD/INFE Toolkit for Measuring Financial Literacy and Financial Inclusion. Available from: https://www.oecd.org/ financial/education/2018-INFE-FinLit-Measurement-Toolkit.pdf.
- [Background] Hoge GL, Stylianou AM, Hetling A, Postmus JL. Developing and Validating the Scale of Economic Self-Efficacy. J Interpers Violence. 2020 Aug;35(15-16):3011-3033. doi: 10.1177/0886260517706761. Epub 2017 May 3. PMID 29294740
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Kaittila A, Isoniemi H, Viitasalo K, Moisio M, Raijas A, Toikka E, Tuominen J, Hakovirta M. A Pilot Randomized Controlled Trial of Intervention for Social Work Clients with Children Facing Complex Financial Problems in Finland (FinSoc): A Study Protocol. J Evid Based Soc Work (2019). 2024 Jan 2;21(1):32-49. doi: 10.1080/26408066.2023.2257174. Epub 2023 Sep 15. PMID 37712670